CLINICAL TRIAL: NCT06717282
Title: Evaluation of a Contextual, Behavioral, and Cognitive-based Program to Improve Ophthalmic Compliance in Children and Adolescents with Special Needs
Brief Title: Evaluation of a Program to Enhance Ophthalmic Compliance in Children and Adolescents with Special Needs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202410102RINB
Record Dates: First submitted 2024-12-01; First posted 2024-12-04 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-11

CONDITIONS: Visual Rehabilitation; Visual Impairment, Autism Spectrum Disorder, Developmental Disabilities, Intellectual Disability, Behavioral Symptoms
Keywords: Visual rehabilitation, Special need, Compliance, Ophthalmic examination
MeSH Terms: conditions — Vision Disorders; Autism Spectrum Disorder; Developmental Disabilities; Intellectual Disability; Behavioral Symptoms; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention to improve ophthalmic compliance (Experimental)
  Interventions: Behavioral: visual rehabilitation for ophthalmic compliance; Behavioral: Using contextual, behavioral, and cognitive-based stragegies to develop training programs

INTERVENTIONS:
Behavioral: visual rehabilitation for ophthalmic compliance — contextual, behavioral, and cognitive-based program for ophthalmic compliance
Behavioral: Using contextual, behavioral, and cognitive-based stragegies to develop training programs — Key Features of the Intervention:
  1. Contextual Adaptation: Participants practice ophthalmic examination procedures in a simulated clinical environment to familiarize themselves with real-world conditions.
  2. Behavioral Strategies: Positive reinforcement, such as rewards (snacks, toys, or videos), is used to encourage participation and cooperation during sessions.
  3. Cognitive Support: Animated materials and interactive exercises are employed to teach the concepts required for visual tests, with take-home tasks for generalization.
  4. Individualized Goals: Individualized training plans and objectives are established collaboratively with caregivers based on participants' cognitive and behavioral profiles.
  Duration and Frequency:
  Six sessions, each lasting one hour, are conducted biweekly, with flexibility based on caregiver availability.

SUMMARY:
The goal of this clinical trial is to learn about the effects of the structured program incorporating contextual, behavioral, and cognitive strategies to improve compliance of children and adolescents with special needs during examinations in specialized or general ophthalmic settings.

The main question it aims to answer is:

"Does this structured program increase ophthalmic examination compliance in children and adolescents with special needs?"

Participants will:

1. Attend six individualized training sessions (one session every two weeks, each lasting one hour)
2. Engage in activities to practice and enhance cooperation during ophthalmic examination
3. Undergo pre- and post-program assessments to measure visal function, behavioral adaptation, and other intervention outcomes.

DETAILED DESCRIPTION:
This study investigates the effectiveness of a contextual, behavioral, and cognitive-based intervention program designed to enhance ophthalmic compliance in children and adolescents with special needs. The program includes six individualized training sessions conducted by occupational therapists with expertise in vision rehabilitation. These sessions integrate environmental adaptation, positive reinforcement, and cognitive strategies to improve the participants' cooperation during ophthalmic examinations.

Intervention Overview:

1. Training Sessions: Each participant will attend six one-on-one sessions over three months, with each session lasting one hour. The frequency of sessions is adjustable but generally follows a biweekly schedule.
2. Structured Strategies: The intervention incorporates contextual strategies (e.g., simulating clinic environments), behavioral reinforcement (e.g., use of rewards), and cognitive tools (e.g., animated instructions) to facilitate learning and generalization of ophthalmic procedures.
3. Parental Involvement: Parents will be engaged throughout the intervention to ensure continuity of training at home.

Quality assurance plan :

1. Regular site monitoring and auditing will be conducted to maintain data quality and protocol adherence.
2. Systematic checks will compare collected data against predefined ranges and consistency rules, ensuring reliability.
3. Missing data will be addressed using standard imputation techniques or sensitivity analyses, ensuring robustness of the results.

Sample Size Assessment:

The study includes a planned sample size of 50 participants, which is deemed sufficient to detect significant changes in primary outcomes with appropriate statistical power.

Analysis Plan:

Primary and secondary outcomes will be assessed using appropriate statistical methods to measure changes in compliance, visual function, and behavior after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 2 and 18 years.
2. Diagnosed with or suspected of having autism spectrum disorder, developmental delay, or intellectual disability.
3. Experiencing difficulties cooperating with routine ophthalmologic examinations in general medical facilities due to cognitive, behavioral, or emotional challenges.

Exclusion Criteria:

* Children and adolescents with developmental delays or disabilities who are capable of undergoing routine vision screenings during regular ophthalmologic visits or school health check-ups.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-21 (Estimated)

PRIMARY OUTCOMES:
Visual Function Battery for Children with Special Needs | 6 months
  Evaluating the multiple visual function of children and adolescent with special needs
Near Detection Scale | 6 months
  The visual acuity assessment tool has a minimum score of 0 and a maximum score of 18. Higher scores indicate better visual acuity.
Functional Vision Questionnaire | 6 months
  Measure visual function and functional vision. The assessment scale has a maximum score of 140 and a minimum score of 28. Higher scores indicate better performance.
Ophthalmic Visit Adaptation Questionnaire | 6 months
  A self-developed scale was designed to evaluate children and adolescents with special needs who experience difficulties in ophthalmic visits. The scale consists of 24 items, rated on a 5-point Likert scale, with a total score of 120. Higher scores indicate greater difficulty in compliance and stability.
Goal Attainment Scale | 6 months
  Quantifying individual goals through discussions with the primary caregiver or the individual themselves after intervention is a highly personalized assessment approach that effectively reflects individual needs.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Occupational Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No